CLINICAL TRIAL: NCT07022691
Title: The Association Between Abdominal Obesity, Gluteal Muscles Strength and Endurance in Young and Middle-aged Adults.
Status: Active, not recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, shady sameh zekry, demonstrator, Cairo University
Other Study IDs: 012/005032
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Obesity in Young and Middle Aged Adults; Gluteal Muscles Strength and Endurance
Keywords: Gluteal Muscles Strength and Endurance,Abdominal Obesity in Young and Middle aged Adults

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: abdominally obese group.: participants will be chosen according to inclusive criteria. The sample size will be calculated depending on pilot study by power analysis (G power).
  Group A: abdominally obese group. Group B: non-abdominally obese group.
  Inclusion Criteria:
  Asymptomatic participants of both sexes with age ranges between 18-50 years. The age range of the participants will be chosen since it corresponds to an economically active group in whom movement disorders can greatly impact function and work. Additionally, individuals over 60 years of age may have reduced muscle mass and function (Artaud et al., 2016).
  Participants with a sedentary lifestyle.
  Exclusion Criteria:
  Pregnancy. an orthopedic disease of the lower limbs. paresthesia or weakness in the lower limb. surgery in the previous years. any other medical conditions affecting lower limb muscle function will be excluded.
  Smokers. Participants who can't do the tests.
  Menopause. BMI more than 30 kg/m2.
  Interventions: Device: Lafayette dynamometer:
- Group B: non-abdominally obese group.: participants will be chosen according to inclusive criteria. The sample size will be calculated depending on pilot study by power analysis (G power).
  Group A: abdominally obese group. Group B: non-abdominally obese group.
  Inclusion Criteria:
  Asymptomatic participants of both sexes with age ranges between 18-50 years. The age range of the participants will be chosen since it corresponds to an economically active group in whom movement disorders can greatly impact function and work. Additionally, individuals over 60 years of age may have reduced muscle mass and function (Artaud et al., 2016).
  Participants with a sedentary lifestyle.
  Exclusion Criteria:
  Pregnancy. an orthopedic disease of the lower limbs. paresthesia or weakness in the lower limb. surgery in the previous years. any other medical conditions affecting lower limb muscle function will be excluded.
  Smokers. Participants who can't do the tests.
  Menopause. BMI more than 30 kg/m2.
  Interventions: Device: Lafayette dynamometer:

INTERVENTIONS:
Device: Lafayette dynamometer: — Lafayette dynamometer will be used for assessment of muscle strength Flexible tape measurement will be used for assessment of WC and hip circumference.

SUMMARY:
to investigate association between abdominal obesity, gluteal muscles strength and endurance in young and middle-aged adults.

DETAILED DESCRIPTION:
participants will be chosen according to inclusive criteria. The sample size will be calculated depending on pilot study by power analysis (G power).

Group A: abdominally obese group. Group B: non-abdominally obese group. The randomization will be performed by computerized randomization. Assessors will be blinded to the groups of the subjects.

Scales and Instrumentation for assessment:

The following instruments will be used as:

Lafayette dynamometer will be used for assessment of muscle strength. Flexible tape measurement will be used for assessment of WC and hip circumference.

All participants will be assessed once. Waist circumference (centimeters) will be determined using a flexible metric tape at the midpoint between the iliac crest and last rib. The participant remained standing with arms alongside the body and the trunk free of clothing. The measurement will be performed with the abdomen relaxed at the end of expiration (Banks et al., 2006).

Men Waist circumference ≥ 102 cm and women Waist circumference ≥ 88 cm (National Heart, Lung, and Blood Institute.2024).

Waist-Hip Ratio measurement:

To measure the waist-to-hip ratio (WHR), first locate the natural waistline, which is typically just above the belly button, and measure its circumference using a tape measure. Then, measure the circumference of the hips at their widest point. Calculate the WHR by dividing the waist circumference by the hip circumference. For example, if your waist measures 80 cm and your hips measure 100 cm, your WHR would be 0.80 (80/100) (World Health Organization, 2008). This ratio will help assess fat distribution and potential health risks, with higher values indicating a greater risk of cardiovascular diseases and other health issues (American Heart Association, 2019).

Familiarization session as it is a critical component in ensuring accurate and reliable results in physical assessments. During this session, participants are introduced to the specific tests and procedures they will undergo, allowing them to become comfortable with the testing environment and equipment. This process typically involves a brief overview of each test, including proper technique, safety measures, and the goals of the assessment. Participants may perform practice trials to get accustomed to the movements and protocols, which helps reduce anxiety and improve performance consistency. Additionally, the familiarization session will allow the assessor to address any questions or concerns, ensuring that participants understand the expectations and can execute the tests effectively. By providing a clear understanding and practice opportunities, the familiarization session will help to minimize variability and enhance the accuracy of the subsequent strength and endurance measurements.

Utilizing a blind assessor for testing muscle strength and endurance will be a crucial strategy to minimize bias and ensure the objectivity of the assessment process. A blind assessor is one who conducts the evaluation without prior knowledge of the participant's identity or their previous performance metrics. This approach helps eliminate any unconscious biases or preconceived expectations that might influence the assessment outcome. By keeping the assessor unaware of such details, the focus remains solely on the participant's current performance, leading to more accurate and fair measurements of muscle strength and endurance. This method not only upholds the integrity of the testing process but also enhances the reliability of the results, as it reduces the potential for subjective interpretation and ensures that all participants are evaluated under the same standardized conditions.

Measuring the strength of the gluteus maximus using a handheld dynamometer is a practical approach for assessing lower body muscle strength, particularly in rehabilitation and sports settings. Here's a guide on how to perform this measurement.

Measurement Procedure

1. Positioning the Subject:

o Prone Position: Have the subject lie face down on a table or mat with their legs extended and feet hanging off the end. This position ensures that the gluteus maximus is isolated and can be effectively tested (Hegedus et al., 2012).

Setting Up the Dynamometer:

* Handheld Dynamometer: Use a handheld dynamometer, such as the dynamometer (Nicholas Manual Muscle Tester, Lafayette Instrument Company, Lafayette, Indiana, USA). Dynamometer should be calibrated and zeroed before use.
* Placement: For the prone position, place the dynamometer on the posterior aspect of the thigh, just above the knee joint (Mathur & Singh, 2011).

Performing the Test:

• Prone Position Test: Ask the subject to extend their hip (lift the thigh upward) against resistance applied by the dynamometer. The tester should apply a consistent, opposing force while the subject exerts maximal effort. (Moffroid & Kottke, 1976).

Recording Measurements:

* Instruct the subject to perform the movement slowly and steadily. The peak force exerted by the subject should be recorded. Typically, a few trials are performed, and the highest value is used for analysis (Bohannon, 2005).
* Subject will perform the movement three trials and the peak one will be chosen.

ELIGIBILITY:
Inclusion Criteria:

Asymptomatic participants of both sexes with age ranges between 18-50 years. The age range of the participants will be chosen since it corresponds to an economically active group in whom movement disorders can greatly impact function and work. Additionally, individuals over 60 years of age may have reduced muscle mass and function (Artaud et al., 2016).

Participants with a sedentary lifestyle. -

Exclusion Criteria:

Pregnancy. an orthopedic disease of the lower limbs. paresthesia or weakness in the lower limb. surgery in the previous years. any other medical conditions affecting lower limb muscle function will be excluded.

Smokers. Participants who can't do the tests. Menopause. more than 30 kg/m2.

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The purpose of the study will be to investigate the association between abdominal obesity, gluteal muscles strength and endurance in young and middle-aged adults.
  Design of the study: cross sectional study
  Subjects of the study:
  participants will be chosen according to inclusive criteria. The sample size will be calculated depending on pilot study by power analysis (G power).
  Group A: abdominally obese group. Group B: non-abdominally obese group.
  Inclusion Criteria:
  Asymptomatic participants of both sexes with age ranges between 18-50 years. The age range of the participants wilyears. The age range of the participants will be chosen since it corresponds to an economically active group in whom movement disorders can greatly impact function and work. Additionally, individuals over 60 years of age may have reduced muscle mass and function Participants with a sedentary lifestyle.
  Exclusion Criteria:
  Pregnancy. an orthopedic disease of the lower limbs.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
assessment of WC and hip circumference. | 1 minute
  Flexible tape measurement will be used
assessment of muscle strength. | 3 minutes
  Lafayette dynamometer will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No